CLINICAL TRIAL: NCT06264011
Title: Discrimination and Religious Experiences of Adult Muslimahs in Salaat
Acronym: DREAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023B0044
Record Dates: First submitted 2023-10-30; First posted 2024-02-16 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Stress, Psychological; Control
MeSH Terms: conditions — Stress, Psychological | interventions — Faith Healing

STUDY DESIGN:
Intervention Model Description: There is one intervention (i.e., the prayer condition) and one control condition (i.e., the counting condition).
Who Masked: Investigator
Masking Description: This study uses a cross-sectional, repeated measures, crossover design. All participants will complete both conditions of the study but will be randomized to start in either the salaat or counting conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salaat (Experimental): The salaat consists of praying the Duha prayer, an optional superogatory prayer that typically occurs in the early morning, to control for differences in timing and duration of prayer. The Duha is completed between the dawn and noon prayers and consists of four cycles of prayer as well as Qur'an recitation and supplication throughout the four positions. The salaat condition includes four cycles with four different positions during each cycle (standing with bowing at a 90-degree angle with both hands covering the knees, standing again briefly with arms at the sides, prostrating with forehead, hands, knees, and feet touching the ground, followed by sitting with knees bent under the torso, prostrating, and sitting again).
  Interventions: Behavioral: Salaat
- Counting (Sham Comparator): The counting condition will include the same physical component as the salaat condition. This will include 4 cycles of movement through the four different positions (i.e., standing, bowing at a 90-degree angle with both hands covering the knees, standing again briefly with arms at the sides, prostrating with forehead, hands, knees, and feet touching the ground, followed by sitting with knees bent under the torso, prostrating, and a final sitting position in cycles two and four. The counting condition will include replacing Qur'anic recitation and subsequent supplications throughout the prayer by counting "one one-thousand, two one-thousand, three one-thousand, etc." throughout the duration of time typically required to perform the full salaat.
  Interventions: Other: Sham comparator

INTERVENTIONS:
Behavioral: Salaat — While Muslims perform mandatory salaat (prayer) 5 times daily, the Duha salaat is an optional daily prayer consisting of 4 cycles of standing, bowing, standing again, prostrating, kneeling, and prostrating again. Research has shown that salaat may influence physiological relaxation.
  Other Names: salaah; Prayer
  Arms: Salaat
Other: Sham comparator — Participants will count while mimicking the movements of the Duhaa salaat. This is a no-prayer condition in which the recitation of Qur'an is omitted for the sake of comparison.
  Other Names: Counting condition; Sham condition
  Arms: Counting

SUMMARY:
This goal of this clinical trial is to examine the effects of the Muslim prayer (salaat) on physiological arousal among Muslim women. This study aims to measure EEG and HRV during the salaat performance among Muslim women. Using EEG as a measure of physiological relaxation, HRV will be utilized as a measure of stress experienced by Muslim women whose prayer have been understudied in research on the salaat. Thus, the main questions it aims to answer are 1) whether salaat performed by Muslim women influences physiological relaxation similar to what is seen by men, and 2) Evaluate health-related correlates of perceived discrimination among Muslim women.

Participants will complete 15 questionnaires. Participants will be connected to a Heart Rate Variability (HRV) monitor as well as a 32-electrode EEG cap. After the baseline data are obtained, all participants will complete both conditions (salaat and counting) but the order of participation in conditions will be randomly assigned. The resting period will again occur between conditions and at the end of the second condition.

All participants will pray the Duha prayer, an optional superogatory prayer that typically occurs in the early morning, to control for differences in timing and duration of prayer. The Duha is completed between the dawn and noon prayers and consists of four cycles of prayer as well as Qur'an recitation and supplication throughout the four positions. The salaat condition includes four cycles with four different positions during each cycle (standing with bowing at a 90-degree angle with both hands covering the knees, standing again briefly with arms at the sides, prostrating with forehead, hands, knees, and feet touching the ground, followed by sitting with knees bent under the torso, prostrating, and sitting again). The counting condition will include the same physical component as the salaat condition. This will include 4 cycles of movement through the four different positions (i.e., standing, bowing at a 90-degree angle with both hands covering the knees, standing again briefly with arms at the sides, prostrating with forehead, hands, knees, and feet touching the ground, followed by sitting with knees bent under the torso, prostrating, and a final sitting position in cycles two and four (see Figure 2)). Apart from not including the final sitting position, cycles one and three are identical to cycles two and four (see Figure 2). The counting condition will include replacing Qur'anic recitation and subsequent supplications throughout the prayer by counting "one one-thousand, two one-thousand, three one-thousand, etc." throughout the duration of time typically required to perform the full salaat. During the standing position, counting can last for approximately 30-60 seconds in line with the previous study by Doufesh and colleagues (2012). Thus, the first three cycles of prayer will require approximately 77 seconds each while the final cycle will require around 97 seconds based on the estimates by Doufesh and colleagues (2012), for a total of approximately five and a half minutes. To ensure that participant duration during the counting condition is, on average, equivalent to the salaat condition, an audio recording will be provided with counting aloud during each position. The duration of the counting in the audio recording will be an average of the duration of each position as found in Doufesh and colleagues (2012). A bell sound will be used to indicate when participants should change to the next position. After performance of each condition, participants will return to a comfortable seated position. Participants will complete a questionnaire to rate their mental focus in the condition. Blood pressure will be measured at the end of each condition. While at rest, assessment of blood pressure, HRV, and EEG will be obtained from participants for 5 minutes between each condition and at the end of the study.

DETAILED DESCRIPTION:
Over the past 30 years, research has increasingly focused on the impact of religious practices on stress reduction. The Islamic prayer (salaat) is a mind-body practice consisting of a movement component and a meditative component. Although Weigand and colleagues (2004) and others (Archour & Roslan, 2014; Archour, Muhamad, Syihab, Mohd, & Mohd, 2021) have demonstrated robust negative associations between the practice of the Muslim prayer form (salaat) and anxiety. More recently, Doufesh and colleagues (2012; 2014; 2018) have examined the effect of salaat on central nervous system (CNS) and cardiovascular functioning. These studies have demonstrated improved physiological relaxation as reflected in increased alpha wave activity and high frequency heart rate variability (HF-HRV) among men. To date, existing studies that have focused on the relationships of salaat with anxiety and cardiovascular functioning have been mostly single group, observational designs. The only prior study with a control condition utilized a resting state comparison group rather than a true sham condition (Gao et al., 2019). Also, past studies have focused almost exclusively on Muslim men. Finally, research has documented the harmful effects of discrimination on automatic nervous system (ANS) functioning on racial and ethnic minorities (Nikolova, Tzacheva, & Vodenitcharov, 2011). However, a paucity of research has examined the relationship of salaat and ANS functioning among Muslim women or Muslimahs reporting experiences of perceived discrimination. This is particularly important as discrimination reported by Muslim women is positively associated with their visibility, e.g., greater adherence to Islamic practices such as the traditional headscarf and wearing loose clothing in public spaces is associated with increased experience of discrimination (Ali, Elsayed, Elahi, Zia, & Awaad, 2022). Thus, this study was designed to evaluate the influence of the recitation component of salaat on ANS functioning among visible Muslim women using a sham control condition. In addition, this study will explore the degree to which perceived discrimination is associated with physiological markers of stress and with health behaviors among Muslim women. Thus, this study aims to replicate and expand upon previous research demonstrating that alpha wave activity during EEG recordings can be found during the salaat.

ELIGIBILITY:
Inclusion Criteria:

* Adult Muslim women;
* Ages 18-55;
* Being ability to complete the salaat without assistance.

Exclusion Criteria:

* Being currently pregnant;
* Being post-menopausal or having a lack of regular menstrual cycles;
* Reporting a current neurological or psychological disorder;
* Receiving a score of greater than or equal to 9 on the Patient Health Questionnaire-9 (PHQ-9);
* Being unable or unwilling to follow the requirements of the study protocol;
* Being unwilling or unable to complete the morning salaat unassisted;
* Being unable or unwilling to provide written informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants must be Muslim women.
Enrollment: 42 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Relative power alpha | Relative power alpha will be assessed beginning five minutes prior to the first condition (salaat/sham condition) and will continue through the study until five minutes after the second condition, for a total duration of around 30-45 minutes.
  Electroencephalography (EEG) is an indicator of relaxation. EEG, a measure of electrical brain activity in various regions of the brain (Luck, 2014), can be used to demonstrate changes in CNS activity attributable to relaxation (Jacobs & Friedman, 2004). During performance of the salaat, HRV may be measured in frequency bands of low frequency (LF) ranging from about 0.04 - 0.15 Hz and high frequency (HF) ranging from about 0.15-0.40 Hz.
High frequency heart rate variability (HF-HRV) | HF-HRV will be assessed beginning five minutes prior to the first condition (salaat/sham condition) and will continue through the study until five minutes after the second condition, for a total duration of around 30-45 minutes.
  Using a heart-rate variability monitor, low sympathetic nervous system activity and higher peripheral nervous system (PNS) activity is measured as high frequency heart rate variability (HF-HRV).
  Using a heart-rate variability monitor, low sympathetic nervous system activity and higher PNS activity is measured as high frequency heart rate variability (HF-HRV).
The Body Perception Questionnaire Body Awareness Very Short Form (BPQ-VSF) | IPAQ-SF will be measured only during the baseline, a single time-point prior to the intervention.
  The Body Perception Questionnaire Body Awareness Very Short Form BPQ-VSF is a 12-item self-report measure adapted from the shortened version of the 26-item BPQ-SF to assess Autonomic nervous system function using a single factor of body awareness (Kolacz et al., 2018). Categorical omega was calculated for internal consistency yielding .91 for the full scale (Cabrera et al., 2018). Test-retest reliability was .97 (Cabrera et al., 2018). Scores range from 12 - 60 with higher scores indicating greater ANS functioning.

SECONDARY OUTCOMES:
The SF 36-Item Health Survey (SF-36) | The SF-36 will be measured only during the baseline, a single time-point prior to the intervention.
  The 36-Item Health Survey short form (SF-36) is a 36-item self-report measure assessing health-related quality of life in eight domains: physical functioning, role limitations due to physical health problems, role limitations due to personal or emotional problems, general mental health, bodily pain, social functioning, general health perceptions, and energy/fatigue. The scale also yields two component scores: a mental component summary score (MCS) and a physical component summary (PCS) score (Hays, Sherbourne, & Mazel, 1993). The MCS and PCS scores will be utilized in this study to reflect generic quality of life in the emotional (MCS) and physical (PCS) domains. Possible scores of the components range from 0 to 100, with higher scores indicating more favorable health state. Cronbach's alpha for the current study was 0.87 for both the PCS and MCS domains.
Modified International Physical Activity Questionnaire - Short Form (IPAQ-SF) | IPAQ-SF will be measured only during the baseline, a single time-point prior to the intervention.
  The Modified International Physical Activity Questionnaire - Short Form (IPAQ-SF; Craig et al., 2003) is an 8-item self-report measure that assesses physical activity and inactivity during the previous seven days. The IPAQ-SF demonstrates acceptable criterion validity (pooled ρ = .30), and respondents report the number of days, hours per day, and minutes per day in the last seven days that they engaged in vigorous exercise, moderate exercise, walking, and sitting. Five factors are scored including total physical activity, walking, moderate activity, vigorous activity, and sitting (Lee, Macfarlane, Lam, & Stewart, 2011).
Health Care Discrimination Scale (HCDS; Martin, 2015) | The HCDS will be measured only during the baseline, a single time-point prior to the intervention.
  The Health Care Discrimination Scale (HCDS) is a 15-item scale comprised of two subscales: the health care cultural safety subscale (HCCS), and the healthcare provider addressed Muslim-specific care needs of patient and family subscale (HCPF) (Martin, 2015). Possible scores for the total measure range from 0 - 48. The range of scores for the HCCS and HCPF subscales are both 0 - 24. Cronbach's alpha for the overall HCDS was α = .78 while the HCCS and HCPF subscales demonstrated reliability estimates of α = .87 and α = .66 respectively (Martin, 2015).
Perceived Religious Discrimination Scale (PRDS; Rippy & Newman, 2008) | The PRDS will be measured only during the baseline, a single time-point prior to the intervention.
  The Perceived Religious Discrimination Scale (PRDS) is a 36-item self-report measure of perceived discrimination based on religious identity. Participants respond to items on a 5-point Likert scale from zero (never) to four (very frequently). All items can be summed for a total score. Additionally, there are three subscales that can be calculated: Racial Prejudice and Stigmatization (RPS), Bicultural Identification (BI), and Racist Environment (RE). The PRDS exhibits high internal reliability for the total score (Cronbach's α = .92) and for the three subscales: RPS (α = .91), BI (α = .84), and RE (α = .87) (Rippy & Newman, 2008). Possible scores for the total measure range from 0 - 132. The range of scores for the RPS, BI, and RE subscales are 0 - 88, 0 - 20, and 0 - 24, respectively.
The Internalized Islamophobia Scale | The IIS will be measured only during the baseline, a single time-point prior to the intervention.
  The Internalized Islamophobia Scale (IIS) was adapted from the Appropriated Racial Oppression Scale for use with Muslim individuals (AROS; Campon R. R., & Carter, R.T. 2015). After removal of the American Standards of Beauty subscale, the original 24-item scale was reduced to 15 items consisting of 3 of the 4 original factors: emotional responses (ER), devaluation of one's own group (DG), and patterns of thinking (PT) (Campon R. R., & Carter, R.T. 2015). Cronbach's alpha internal reliability for the AROS was α=.83 for ER subscale, α=.86 for DG subscale, and α=.70 for the PT subscale (Campon R. R., & Carter, R.T. 2015). Possible scores for the total measure range from 15 - 105. The range of scores for the ER, DG, and PT subscales are 6 - 42, 6 - 42, and 3 - 21, respectively.
Muslim Identification Scale (MIS; Verkuyten, 2007) | The MIS will be measured only during the baseline, a single time-point prior to the intervention.
  The Muslim Identification Scale (MIS) is a 6-item self-report measure of the degree to which individuals who categorize themselves as Muslim identify with their own faith, rated on a 5-point likert scale (strongly disagree to strongly agree). This 6-item scale measures several aspects of religious identification such as importance of faith, religiosity, identification with other Muslims, and mosque or masjid attendance. A single index is calculated for each respondent by adding his or her responses to the six items. The Muslim Identity Scale has demonstrated strong internal consistency with a reported Cronbach's α of .95 (Verkuyten, 2007). Possible scores for the total scale range from 6 - 30.
Brief Religious COPE | The Brief RCOPE will be measured only during the baseline, a single time-point prior to the intervention.
  The Brief Religious Cope (Brief RCOPE) is a 14-item measure assessing religious coping in the face of major life stressors. The Brief RCOPE has two subscales: positive religious coping (PRC) and negative religious coping (NRC). While positive religious coping reflects a constructive relationship with a transcendental force, connectedness with others, and a compassionate worldview, negative religious coping reflects spiritual struggles with oneself, others, and with the divine. The NRC subscale has emerged as a robust predictor of health-related outcomes (Pargament, Feuille, & Burdzy, 2011).
Salaat Frequency Scale | The SFS will be measured only during the baseline, a single time-point prior to the intervention.
  The Salaat Frequency Scale (SFS) is a single item measure of the frequency of salaat performance. Possible scores for the total scale range from 0 to 4. The Salaat Quality Scale is a measure of mindful engagement in salaat according to Islamic goals of obtaining khushu (sincerity and humility), through Ihsan (awareness of God), and taqwa (God consciousness). Possible scores for the scale range from 0 to 32.
The Salaat Index | The Salaat index will be measured only during the baseline, a single time-point prior to the intervention.
  The Salaat Index was adapted from Toylamat and Moradi's Hijab Index (2011) and is a calculation of salaat performance that includes both a qualitative and quantitative component. The Salaat Index is calculated by multiplying Salaat Frequency Scale and Salaat Quality Scale to obtain both qualitative and quantitative measures of the prayer. Possible scores for the total scale range from 0 to 128.
Hijab Frequency Scale | The Hijab Frequency scale will be measured only during the baseline, a single time-point prior to the intervention.
  The Hijab Frequency Scale is a measure of how often participants wear the hijab. Possible scores for the total scale range from 0 to 4. The Hijab Conservativeness Scale ranges from 1 to 8 and measures the extent to which participants wear the traditional Islamic hijab. The Hijab Index is a calculation of hijab use that includes both a qualitative and quantitative component. The Hijab Index is calculated by multiplying hijab conservativeness and hijab frequency to obtain both a qualitative and quantitative measure of hijab (Toylamat & Moradi, 2011). Possible scores for the total scale range from 0 to 32.

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Emery, PhD, Principal Investigator — Professor Emeritus
Locations (1):
- The Ohio State University, Columbus, Ohio, United States